CLINICAL TRIAL: NCT00442143
Title: Treatment of Severe Limb Ischemia With Autologous Bonemarrow Derived Mononuclear Cells
Acronym: DANCELL-CLI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 024
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2007-03

CONDITIONS: Ischemia
Keywords: CLI; PAOD; Severe lower limb ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stem cell implantation

SUMMARY:
The aim of the study is to investigate whether implantation of autologous bone marrow derived stem cells in ishemics limbs will improve vascularization

DETAILED DESCRIPTION:
10 patients with severe lower limb ischemia will be included in this pilote trial.

Bonemarrow aspiration will be performed and and the monocuclear cells isolated an injected into the gastrocnemius.

The patiens are followed for 4 months. Were trancutaneous oxygenpressure, ankel and toe blood pressure is measured.

ELIGIBILITY:
Inclusion Criteria:

* Ankle blood pressure < 70 mmgHG
* Either pain at rest and/or ischemic wound
* No possible surgical treatment

Exclusion Criteria:

* Infection
* Malignant disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous oxygen pressure
1st toe blood pressure (strain gauge)
Ankle blood pressure
Wound healing
Pain

SECONDARY OUTCOMES:
amputation
Infection

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Kassem, MD, Principal Investigator — Department of endocrinology M, Odense University Hospital
Locations (1):
- Department of endocrinology M, Odense University Hospital, Odense, Denmark